CLINICAL TRIAL: NCT05614583
Title: Multidisciplinary Digital Therapeutics of Patellofemoral Pain Syndrome Versus Usual Care, a Randomized Controlled Pilot Study
Brief Title: Multidisciplinary Digital Therapeutics of Patellofemoral Pain Syndrome Versus Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EverEx Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-ETH-01K-CTP-01
Record Dates: First submitted 2022-10-30; First posted 2022-11-14 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Single site, randomized controlled trial research study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MORT-PFPS (Experimental): Participants randomly assigned to this arm will use the app, MORT-PFPS.
  Interventions: Device: MORT-PFPS app
- treatment as usual (TAU) (Active Comparator): Participants randomly assigned to this arm will receive their TAU only (no use of the app, MORT-PFPS).
  Interventions: Other: treatment as usual (TAU)

INTERVENTIONS:
Device: MORT-PFPS app — The MORT-PFPS, developed by EverEx, Inc., is designed to provide multidisciplinary rehabilitation treatment, a combination of graded exercise therapy and cognitive behavioural therapy for patients with patellofemoral pain syndrome.
  Arms: MORT-PFPS
Other: treatment as usual (TAU) — In the control group, psychoeducation is delivered and self-exercise is recommended.
  Arms: treatment as usual (TAU)

SUMMARY:
This randomized controlled pilot study will be evaluating an app, MORT-PFPS app (ETH-01K), owned by EverEx, Inc., to examine safety and effectiveness in individuals with patellofemoral pain syndrome.

DETAILED DESCRIPTION:
This randomized controlled pilot study will enroll 40 participants, where half will be randomly assigned to the app, MORT-PFPS (n = 20), and half will be assigned to treatment as usual (TAU) (n = 20), to examine safety and effectiveness in individuals with patellofemoral pain syndrome. All subjects will be followed up in the study for a total of 12 weeks, 8-week courses of treatment with additional 4-week observation. The app provides multidisciplinary rehabilitation treatment, a combination of graded exercise therapy and cognitive behavioural therapy for patients with patellofemoral pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 19 and <50 years of age
* Patients who have a history of anterior knee pain in one or both knees, persisting for longer than 3months but not longer than 2 years
* Patients who have pain provoked by squatting
* Patients who have pain provoked by 2 or more following activities

  1. long sitting
  2. cycling
  3. running
  4. going up or down stairs
  5. kneeling
  6. compression of the patella
  7. palpation of the patellar facets
* Patients who signed a written informed consent form

Exclusion Criteria:

* Patients with osteoarthritis which scored 2 or higher grade of the Kellgren-Lawrence scale
* Patients who have a history of knee pathologies or injuries (fracture, tendon injury, cartilage injury, or patella dislocation)
* Patients who had previous knee surgeries
* Patients who have patellar tendinopathy
* Patients who have Osgood-Schlatter disease, or other defined pathological conditions of the knee
* Patients who are pregnant or breastfeeding
* Patients who are using anti-inflammatory medication
* Patients with known substance/alcohol use disorders
* Patients with known somatic symptom and related disorders
* Patients who are not able to participate in an exercise or strengthening program

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Usual pain severity assessed by the Numeric Rating Scale (NRS ) | 8 weeks
  The primary outcome being measure is differences in usual pain severity between groups after the intervention. NRS score was measured from 0 (no pain) to 10 (worst pain imaginable).
Global rating of perceived recovery | 8 weeks
  The primary outcome being measure is differences in global rating of perceived recovery between groups after the intervention. Global rating of perceived recovery score was measured from 1 (very bad) to 7 (very good).
Functional disability assessed by the Kujala Patellofemoral Scale | 8 weeks
  The primary outcome being measure is differences in functional disability between groups after the intervention. Kujala Patellofemoral Scale, also known as Anterior Knee Pain Scale, is a patient reported assessment of patellofemoral pain syndrome-specific functional limitations. It has 13 questions, and total score ranges from 0 to 100 (higher scores meaning better outcomes).

SECONDARY OUTCOMES:
Usual pain severity assessed by the Numeric Rating Scale (NRS) | 4, 12 weeks
  The secondary outcome being measure is differences in usual pain severity between groups at 4 and 12 weeks. NRS score was measured from 0 (no pain) to 10 (worst pain imaginable).
Global rating of perceived recovery | 4, 12 weeks
  The secondary outcome being measure is differences in global rating of perceived recovery between groups at 4 and 12 weeks. Global rating of perceived recovery score was measured from 1 (very bad) to 7 (very good).
Functional disability assessed by the Kujala Patellofemoral Scale | 4, 12 weeks
  The secondary outcome being measure is differences in functional disability between groups at 4 and 12 weeks. Kujala Patellofemoral Scale, also known as Anterior Knee Pain Scale, is a patient reported assessment of patellofemoral pain syndrome-specific functional limitations. It has 13 questions, and total score ranges from 0 to 100 (higher scores meaning better outcomes).
Worst pain severity, pain during specific activities (running, standing up from sitting, going up or down stairs, and sleeping) assessed by the Numeric Rating Scale (NRS) | 4, 8, 12 weeks
  The secondary outcome being measure is differences in worst pain severity, pain during specific activities between groups at 4, 8 and 12 weeks. NRS score was measured from 0 (no pain) to 10 (worst pain imaginable).
Health-related quality of life assessed by EuroQol five-dimensional (EQ-5D) | 4, 8, 12 weeks
  The secondary outcome being measure is differences in health-related quality of life between groups at 4, 8 and 12 weeks. It measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with three possible answers for each dimension (1=no problem, 2=moderate problem, 3=severe problem). The instrument also includes a visual analogue scale, which is numbered from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Changes of Knee strength | 8, 12 weeks
  Flexion and extension strength of knee are measured using a Biodex isokinetic dynamometer (peak torque (Nm) and % decrease in torque).
Changes of hip abductor function | 8, 12 weeks
  Hip abductor function is assessed by knee valgus angle during single leg squat (°).
Changes of usual pain severity, worst pain severity, pain during specific activities (running, standing up from sitting, going up or down stairs, and sleeping), assessed by the Numeric Rating Scale (NRS) | 4, 8, 12 weeks
  The secondary outcome being measure is differences in changes of usual pain severity, worst pain severity, pain during specific activities from baseline to 4, 8, and 12 weeks between groups. NRS score was measured from 0 (no pain) to 10 (worst pain imaginable).
Changes of functional disability assessed by the Kujala Patellofemoral Scale | 4, 8, 12 weeks
  The secondary outcome being measure is differences in changes of functional disability from baseline to 4, 8, and 12 weeks between groups. Kujala Patellofemoral Scale, also known as Anterior Knee Pain Scale, is a patient reported assessment of patellofemoral pain syndrome-specific functional limitations. It has 13 questions, and total score ranges from 0 to 100 (higher scores meaning better outcomes).
Changes of health-related quality of life assessed by EuroQol five-dimensional (EQ-5D) [ Time Frame: 4, 8, 12 weeks ] | 4, 8, 12 weeks
  The secondary outcome being measure is differences in changes of health-related quality of life from baseline to 4, 8, and 12 weeks between groups. It measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with three possible answers for each dimension (1=no problem, 2=moderate problem, 3=severe problem). The instrument also includes a visual analogue scale, which is numbered from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Assessment of mental health symptoms specific to depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | 8, 12 weeks
  Differences in mental health symptoms between groups at 8, 12 weeks. The Patient Health Questionnaire-9 (PHQ-9) total score for the nine items ranges from 0 to 27 (higher scores indicating greater severity of depression).
Assessment of catastrophic thinking measured by Pain Catastrophizing Scale (PCS) | 8, 12 weeks
  Differences in levels of catastrophic thinking between groups at 8, 12 weeks. The Pain Catastrophizing Scale (PCS) is a 13-item scale, with a total range of 0 to 52 (higher scores indicating higher amounts of pain catastrophizing).
Assessment of fear avoidance behaviours measured by Fear-Avoidance Beliefs Questionnaire (FABQ) | 8, 12 weeks
  Differences in fear avoidance behaviours between groups at 8, 12 weeks. The Fear-Avoidance Beliefs Questionnaire (FABQ) is a 16-item scale, with a total range of 0 to 96 (higher scores indicating higher amounts of fear avoidance behaviours).
Use of rescue medication | 4, 8, 12 weeks
  Differences in use of rescue medication between groups at 4, 8, 12 weeks.
Assessment of retention in treatment | 4, 8 weeks
  Differences in retention rates between groups at 4, 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Chong Bum Chang, Dr., Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul Metropolitan Government-Seoul National University Boramae Medical Center, Dongjak, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee S, Yoon C, Choi CH, Park TH, Yang SJ, Cha HR, Kim TW, Park JH, Chang MJ, Chang CB. Efficacy of a Mobile Multidisciplinary Digital Therapeutics App for Patellofemoral Pain: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2025 Oct 17;13:e69627. doi: 10.2196/69627. PMID 41105952